CLINICAL TRIAL: NCT06260137
Title: Comparison of the Effectiveness of the Combination of Rhomboid Intercostal and Sub-serratus Plan Block and Rhomboid Intercostal Block for Postoperative Analgesis in Video-assisted Thoracopic Surgery (VATS)
Brief Title: Comparison of Two Different Methods for Reducing Pain After Lung Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Ferhat Ustuner, Research Assistant Doctor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UludagThorax
Record Dates: First submitted 2024-02-01; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Analgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhomboid İntercostal Block (RIB) (Active Comparator)
  Interventions: Procedure: Rhomboid intercostal block
- Rhomboid intercostal and subserratus plane block (RISS) (Active Comparator)
  Interventions: Procedure: Rhomboid intercostal and subserratus plane block

INTERVENTIONS:
Procedure: Rhomboid intercostal block — Patients will be injected with a local anesthetic drug under the rhomboid intercostal muscle before surgery.
  Arms: Rhomboid İntercostal Block (RIB)
Procedure: Rhomboid intercostal and subserratus plane block — Patients will be injected with a local anesthetic drug under the rhomboid intercostal muscle and the serrates anterior muscle before surgery.
  Arms: Rhomboid intercostal and subserratus plane block (RISS)

SUMMARY:
The goal of this clinical study is to compare the effectiveness of the Rhomboid Intercostal Block and Sub-Servitus plan block and the effectiveness of the Rhomboid intercostal block in patients with video-supported thoracoscopic surgery. The main question it aims to answer is:

Which of these two blocks more effectively reduces the patients' pain?

ELIGIBILITY:
Inclusion Criteria:

* Patients in American Society of Anesthesiologists (ASA) classes I, II and III for whom VATS is planned

Exclusion Criteria:

* Known or suspected local anesthetic allergy
* coagulopathy
* injection site infection
* history of thoracic surgery
* serious neurological or psychiatric disorder
* severe cardiovascular disease
* liver failure
* renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia | first 48 hours postoperatively
  Patients' VAS scores and additional analgesic needs in the first 48 hours will be evaluated. VAS (visual pain scale) corresponds to a value between 0 and 10. A value of 0 means no pain, and a value of 10 is the most severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hastane, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No